CLINICAL TRIAL: NCT06800664
Title: The Impact of an Evidence-Based, Behavioral Cervical Cancer Screening Intervention Among Women Living with HIV in Ghana (HOPE-inG): a Type 2 Hybrid Effectiveness Implementation Trial
Brief Title: Home-based Self-sampling for Cervical Cancer Prevention Education Intervention in Ghana
Acronym: HOPE-inG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Matt Asare, Assistant Professor, Baylor University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1U01CA294757-01 (NIH); 1U01CA294757-01 (NIH)
Record Dates: First submitted 2024-12-12; First posted 2025-01-30 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer Screening; HIV; Self-sampling; Implementation Science; Intervention (Training) Condition; Implementation Strategies
MeSH Terms: interventions — Capacity Building; Control Groups

STUDY DESIGN:
Intervention Model Description: Aim 1: This study uses mixed-method approaches (qualitative and quantitative). Through nominal group techniques (NGT) (qualitative method), the investigators will support engaged stakeholders in selecting, prioritizing, and adapting culturally appropriate implementation support strategies (ISS) for HOPE. Surveys (quantitative method) will be used to evaluate the feasibility, acceptability, and appropriateness of HOPE 2.0 and prioritized/refined ISS.
  Aims 2 & 3: Investigators will conduct a hybrid type2 cluster RCT to evaluate the effectiveness of HOPE 2.0 and the implementation of HOPE 2.0 using bridging factor-focused ISS at secondary health facilities. HIV clinics at four secondary facilities will be cluster-randomized 1:1 in a two-arm trial. WLWH in the Intervention group will receive HOPE 2.0 from providers trained with ISS in implementing to be developed and adopted WLWH in the control group will also receive HOPE 2.0, but from providers who did not receive implementation training
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Health providers and management at IG sites will receive ISS (i.e., management support, capacity-building, and social network support) and training on the HOPE implementation plan
  Interventions: Behavioral: Health providers and management at IG sites will receive ISS (i.e., management support, capacity-building, and social network support) and training on the HOPE implementation plan; Behavioral: Control Group
- Control Group (No Intervention): Providers and management in the control group will not receive any ISS or implementation plan training

INTERVENTIONS:
Behavioral: Health providers and management at IG sites will receive ISS (i.e., management support, capacity-building, and social network support) and training on the HOPE implementation plan — Health providers and management at IG sites will receive ISS (i.e., management support, capacity-building, and social network support) and training on the HOPE implementation plan
  Arms: Intervention Group
Behavioral: Control Group — Providers in the control group will not receive ISS support
  Arms: Intervention Group

SUMMARY:
The investigators propose to develop and/or adapt implementation strategies and a structured implementation plan to translate the HOPE intervention into existing healthcare practice in Ghana.

These "implementation support strategies (ISS)" are implementation strategies relevant to implementation support, which is concerned with moving (implementation) research into (implementation) practice.

The ultimate goal is to facilitate health system adoption and sustainment.

DETAILED DESCRIPTION:
Over 69,000 women living with HIV, (WLWH) in Ghana have a six-fold increased risk of developing cervical cancer and require early and frequent cervical cancer screening (CCS). However, available data in Ghana show that the CCS rate among eligible women is as low as 2.7%, and there is no evidence that WLWH screen at higher rates. In response to the need to increase the uptake of CCS among WLWH, the investigators developed a Home-based self-sampling for cervical cancer Prevention Education (HOPE) intervention. HOPE consists of HPV self-sampling combined with a 3R (Reframing, Reprioritizing, and Reforming) communication model for promoting CCS. In a randomized controlled trial (RCT) in Ghana, the investigators demonstrated that HOPE significantly increased CCS among WLWH (100%) vs routine clinic-based screening (14.64%). Participating women found the self-sampling and 3R communication model acceptable and culturally appropriate. High-impact implementation strategies are needed to integrate and scale up HPV self-sampling into women's healthcare in Ghana. The investigators propose to develop and/or adapt implementation strategies to maximize the success of the HOPE intervention in increasing its health system adoption, patient uptake, and the sustainment of CCS among WLWH. The investigators' proposed hybrid type 2 effectiveness-implementation RCT trial will leverage existing relationships with secondary-level health facilities in Ghana. The investigators will select four secondary-level health facilities with comparable infrastructure and WLWH patient enrollment. Using the Exploration, Preparation, Implementation, and Sustainment (EPIS) framework, the investigators will address the following specific aims.

Aim 1: To develop a culturally appropriate, evidence-based health system implementation plan and provider training content for successful HOPE implementation (Preparation phase). Through nominal group techniques (NGTs), the investigators will support engaged stakeholders in selecting, prioritizing, and adapting culturally appropriate implementation support strategies (ISS) for HOPE. Through NGTs, the investigators will modify HOPE and adopt HOPE 2.0

Aim 2: Assess the effectiveness of the HOPE 2.0 intervention and the success of the implementation plan in a hybrid type 2 trial (Implementation phase). The investigators will conduct a hybrid type 2 effectiveness-implementation RCT to evaluate the impact of implementation strategies. Four HIV secondary-level clinics will be cluster-randomized 1:1 in a two-arm RCT. Healthcare providers in the intervention group (IG, Arm 1) will receive evidence-based training validated in Aim 1. After training, trained providers will recruit WLWH (n = 576) from their HIV facilities and implement HOPE. Providers in the control group (CG, Arm 2) who will not be trained with our ISS materials will recruit WLWH (n = 576) and implement HOPE in their clinics.

Aim 3: Assess the impact of the implementation plan on the sustainment of the HOPE intervention at study sites (Sustainment phase). The investigators will assess the impact of HOPE on WLWH screening behaviors and the impact of strategy material on providers' self-efficacy for implementing HOPE across the study arms.

ELIGIBILITY:
Inclusion Criteria:

General criteria

* ability to give consent per Institutional Review Board stipulations
* residing in the Central Region
* having no medical characteristics that would interfere with the ability to participate fully
* the willingness to participate in this study.

  (a) Healthcare provider eligibility: Inclusion criteria include an individual (no gender restrictions) who
* possesses healthcare qualifications (i.e., patient navigators, physicians, nurses, health facility management),
* works at the HIV health facility at study sites,
* is ≥18 years old. (b) Eligibility for women living with HIV (Patients)
* identified female at birth) who
* are living with HIV between 25 and 65 years old (age consistent with WHO CC screening guidelines)
* have never had CC screening (Pap or HPV test),
* have not had a screening for the past 5 years

Exclusion Criteria:

* Women will be excluded if they are pregnant or have had a hysterectomy.
* WLWH who have a cervix are the main target population to develop the HOPE toolkit.
* Women who are below 25 and those who are above 65 years will be excluded.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Implementation Outcome 1A: HOPE 2.0 Program Adoption | 24 months post-randomization
  The first primary outcome of interest is program adoption, defined as the decision of healthcare management and provider's willingness to use HOPE 2.0 (consisting of self-sampling, 3R model, and patient navigators) and ISS materials in the facilities. Adoption will be measured at at 1, 3-, 6-, 12-, and 24 months post-randomization using a Log sheet.
Implementation Outcome 1B: HOPE 2.0 Program Adoption | 24 months post-randomization
  The first primary outcome of interest is program adoption, defined as the decision of healthcare management and provider's willingness to use HOPE 2.0 (consisting of self-sampling, 3R model, and patient navigators) and ISS materials in the facilities. Adoption will be measured at at 1, 3-, 6-, 12-, and 24 months post-randomization using semi-structured interviews.
Implementation Outcome 1C: HOPE 2.0 Program Adoption | 24 months post-randomization
  The first primary outcome of interest is implementation outcomes of adoption in providers defined as the decision of providers willingness to use HOPE 2.0 (consisting of self-sampling, 3R model, and patient navigators) and ISS materials in the facilities. Adoption will be measured 1, 3, 6- 12- and 24 months post-randomization using Likert Scale surveys.
Implementation Outcome 1D: HOPE 2.0 Program Adoption | 24 months post-randomization
  The first primary outcome of interest is implementation outcomes of adoption in patients, defined as the decision of patients' willingness to use HOPE 2.0 (consisting of self-sampling, 3R model, and patient navigators) and ISS materials in the facilities. Adoption will be measured 1, 3, 6- 12- and 24 months post-randomization. At the patient level, adoption will be measured using a 6 item scale.
Implementation Outcome 2A: HOPE 2.0 Implementation cost | 24 months post-randomization
  The second primary outcome of interest is implementation cost, defined as the total expenses for implementing HOPE 2.0. Cost will be assessed at the health facility and patient levels at 1, 3, 6, 12, and 24 months post-randomization. At both levels, implementation costs will be measured using a cost-tracking database.
Implementation Outcome 2B: HOPE 2.0 Implementation cost | 24 months post-randomization
  The second primary outcome of interest is implementation cost, defined as the total expenses for implementing HOPE 2.0. Cost will be assessed at the patient levels at 1, 3, 6, 12, and 24 months post-randomization using an outpatient cost survey
Implementation Outcome 3A: Fidelity of Implementing HOPE 2.0 | During 24 months post-randomization
  The third primary outcome of interest is Fidelity, defined as the degree to which HOPE 2.0/ISS is implemented as planned in the facilities. Fidelity outcome will be measured at the management level using process evaluation checklists throughout the intervention period.
Implementation Outcome 3B: Fidelity of Implementing HOPE 2.0 | During 24 months post-randomization
  The third primary outcome of interest is Fidelity, defined as the degree to which HOPE 2.0/ISS is implemented as planned in the facilities. Fidelity outcome will be measured at management and provider levels using observations throughout the intervention period.
Implementation Outcome 3C: Fidelity of Implementing HOPE 2.0 | During 24 months post-randomization
  The third primary outcome of interest is Fidelity, defined as the degree to which HOPE 2.0/ISS is implemented as planned in the facilities. Fidelity outcome will be measured at management and provider levels through regular review of log sheets.
Implementation Outcome 3D: Fidelity of Implementing HOPE 2.0 | During 24 months post-randomization
  The third primary outcome of interest is Fidelity, defined as the degree to which HOPE 2.0/ISS is implemented as planned in the facilities. Fidelity outcome will be measured the provider level using a 7 item survey.
Implementation Outcome 4A: HOPE 2.0 Program Penetration in the clinics | 6 months post-randomization
  The fourth primary outcome of interest is Program Penetration, defined as integrating HOPE 2.0/ISS within the clinic facilities. We will assess penetration at management and provider levels using activity log sheets at 1 and 6 months post-randomization.
Implementation Outcome 4B: HOPE 2.0 Program Penetration in the clinics | 6 months post-randomization
  The fourth primary outcome of interest is Program Penetration, defined as integrating HOPE 2.0/ISS within the clinic facilities. We will assess penetration outcomes at management and provider levels using interviews at 1 and 6 months post-randomization.
Implementation Outcome 5A: HOPE 2.0 Sustainment in the facilities | 42 month post-randomization
  The final implementation outcome of interest is sustainability, defined as the extent to which the intervention (HOPE 2.0 and ISS) is integrated within the clinics' routine operations. Sustainability will be measured at the provider and management levels using the Sustainment Measurement System Scale at 12, 24, 36, and 42 months (after a 36-42-month post-trial period) post-randomization.
Implementation Outcome 5B: HOPE 2.0 Sustainment in the facilities | 42 month post-randomization
  The final implementation outcome of interest is sustainability, defined as the extent to which the intervention (HOPE 2.0 and ISS) is integrated within the clinics' routine operations. Sustainability will be measured at the provider and management levels using Interviews at 12, 36, and 42 months post-randomization.

SECONDARY OUTCOMES:
Service Outcome 1A: Program Effectiveness in increase provider self-efficacy | 6 months post-randomization
  The first service outcome of interest is Program Effectiveness, defined as the impact of the ISS on healthcare workers' self-efficacy in implementing HOPE 2.0 within their facilities. Program effectiveness outcomes will be measured at provider and management levels using activity log sheets
Service Outcome 1B: Program Effectiveness in increase provider self-efficacy | 6 months post-randomization
  The first service outcome of interest is Program Effectiveness, defined as the impact of the ISS on healthcare workers' self-efficacy in implementing HOPE 2.0 within their facilities. Program effectiveness outcomes will be measured at provider and management levels using interviews at 1 and 6 months post-randomization.
Service Outcome 1C: Program Effectiveness in increase provider self-efficacy | 6 months post-randomization
  The first service outcome of interest is Program Effectiveness, defined as the impact of the ISS on healthcare workers' self-efficacy in implementing HOPE 2.0 within their facilities. Program effectiveness outcomes will be measured at provider level using a survey to measure the program effectiveness at the providers' level at 1 and 6 months post-randomization.
Service Outcome 2A: Patients' cervical screening uptake | 6 months post-randomization
  The service outcome of interest is screening uptake, defined as the completion and return of a self-sample kit and pap test completion. Screening uptake will be measured at the patients' level using surveys at the 1 month and 6 months post-randomization.
Service Outcome 2B: Patients' cervical screening uptake | 6 months post-randomization
  The service outcome of interest is screening uptake, defined as the completion and return of a self-sample kit and pap test completion. Screening uptake will be measured at the patients' level by verifying the electronic medical records at one month and 6 months post-randomization.
Client Outcome 3A: Patient follow-up treatment. | 12 months post randomization.
  The client outcome is patient treatment follow-up, defined as whether patients with positive results follow up for treatment or not. The outcomes will be measured at the patients' level using surveys at 6 and 12 months post-receiving the test results.
Client Outcome 3B: Patient follow-up treatment. | 12 months post randomization.
  The client outcome is patient treatment follow-up, defined as whether patients with positive results follow up for treatment or not. The outcomes will be measured at the patients' level by verifying the patient clinical records at 6 and 12 months post-receiving the test results
Client Outcome: Patient Satisfaction | 6 months post-randomization
  The client outcome of interest is patient satisfaction, defined as the degree to which patients feel their expectations, needs, and preferences are met by participating in the program. Satisfaction outcomes will be measured at the patients' level by using a satisfaction survey at one post-completing intervention and 6 months after receiving treatment for positive results.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Asare, PhD, Principal Investigator — Baylor University; Dorcas Obiri-Yeboah, PhD, Principal Investigator — University of Cape Coast; Nadia Sam-Agudu, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Cape Coast, Capte Coast, Central Region, Ghana